CLINICAL TRIAL: NCT07350356
Title: Bronchoscopic Role in Early Detection of Endobronchial Tuberculosis in Undiagnosed Suspected Pulmonary Tuberculosis Patients.
Brief Title: Bronchoscopic Role in Early Detection of Endobronchial Tuberculosis in Suspected Pulmonary Tuberculosis Patients.
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MD 203/2023
Record Dates: First submitted 2025-12-20; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Endobronchial Mass; Tuberculosis, Pulmonary
Keywords: Fiberoptic bronchoscopy; Endobronchial TB; Smear negative TB; Suspected PTB
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group 1: PTB with concomitant EBTB, group 2: PTB with no concomitant EBTB.: group 1of 41 patients had positive bronchoscopic findings of PTB with concomitant of EBTB, group 2 of 22 patients had PTB with no concomitant EBTB.
  Interventions: Diagnostic Test: fiberoptic bronchoscopy evaluation of endobronchial features of TB

INTERVENTIONS:
Diagnostic Test: fiberoptic bronchoscopy evaluation of endobronchial features of TB — EBTB was classified into seven subtypes by using the Chung's method: actively caseating, fibrostenotic, oedematous-hyperaemic, tumorous, ulcerative, granular, and the non-specific bronchitic subtype.

SUMMARY:
The aim of the present study is to evaluate the role of bronchoscopy in diagnosis of endobronchial tuberculosis in suspected pulmonary tuberculosis patients whose sputum samples are negative for Ziehl Neelsen stain.

DETAILED DESCRIPTION:
Bronchoscopy plays a major role in identification and diagnosis of EBTB. As a general principal, Bronchoscopy -associated with microbiological testing- must be performed on patients whose CT examination results indicate EBTB.

This study will try to focus on the importance of bronchoscopy in diagnosis of endobronchial tuberculosis among suspected pulmonary tuberculosis patients who undergo fiberoptic bronchoscope after being sputum Ziehl Neelsen negative, scarce sputum and/or persistent consolidation on chest radiograph (CXR).

ELIGIBILITY:
Inclusion Criteria:

* o Adults more than18 years.

  * Accept to participate.
  * Suspected pulmonary tuberculosis patients with three negative sputum samples are smear negative, and/or persistent consolidation on chest radiograph (CXR).

Exclusion Criteria:

* o Patients who refuse to participate in the study.

  * Patients who are sputum Ziehl Neelsen positive.
  * Patients who are diagnosed extrapulmonary tuberculosis.
  * Patients who are not fit for bronchoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients will be recruited from Mansoura chest hospital for pulmonary tuberculosis suspected patients who are smear negative for acid fast bacilli.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
the role of fiberoptic bronchoscopy in sputum smear negative and radiologically suspected pulmonary tuberculosis 63 patients in Mansoura chest hospital, bronchoscopy unit for early detection of endobronchial tuberculosis. | 1 year
  bronchoscopic evaluation of tracheobronchial tree for endobronchial tuberculosis lesions in patients with suspected PTB

SECONDARY OUTCOMES:
The clinical presentation, bronchoscopic characteristics in comparison to radiological characteristics of EBTB, and incidence of EBTB subtypes in pulmonary TB patients | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Heba M Shalaby, MD, Principal Investigator — Ain Shams University, Faculty of medicine
Locations (1):
- Heba Shalaby, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication maybe shared
Supporting Information: Study Protocol, SAP
Time Frame: 1 year
Access Criteria: personal request